CLINICAL TRIAL: NCT02953652
Title: A Phase 2b Open-Label Single Arm Study to Evaluate the Efficacy and Safety of Oral HBI-8000 in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
Brief Title: Efficacy and Safety of Oral HBI-8000 in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HUYABIO International, LLC. (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBI-8000-203
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Peripheral T-Cell Lymphoma (PTCL)
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — HBI-8000

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HBI-8000 (Experimental): Four 10 mg tablets or less twice weekly orally approximately 30 minutes after any regular meal. The treatment will be continuous, with 3-4 days between dosing. Treatment will continue until disease progression in the absence of unacceptable toxicity.
  Interventions: Drug: HBI-8000

INTERVENTIONS:
Drug: HBI-8000 — Orally twice weekly

SUMMARY:
Phase 2b, open-label, non-randomized, single arm study to evaluate the safety, efficacy, and pharmacokinetics of HBI-8000 40 mg BIW in patients with relapsed or refractory PTCL (R/R PTCL).

DETAILED DESCRIPTION:
This is a Phase 2b, open-label, non-randomized, single arm study to evaluate the safety, efficacy, and pharmacokinetics of HBI-8000 40 mg BIW in patients with relapsed or refractory PTCL (R/R PTCL). HBI 8000 will be administered orally approximately 30 minutes after any regular meal twice a week. There will be 3-4 days between dosing. A cycle is defined as consecutive 28 days. HBI-8000 administration will be continued until disease progression or unacceptable toxicities are observed despite appropriate dose reduction or treatment interruption.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis of the following peripheral T-cell lymphoma (PTCL) subtypes as defined by the WHO classification (2008) may be included:

   1. PTCL, NOS
   2. Angioimmunoblastic T-cell lymphoma (AITL)
   3. Anaplastic large-cell lymphoma (ALCL), ALK+
   4. Anaplastic large-cell lymphoma (ALCL), ALK-
   5. Enteropathy-associated T-cell lymphoma (EATL)
   6. Hepatosplenic T-cell lymphoma
   7. Subcutaneous panniculitis-like T-cell lymphoma
2. Patients for whom at least 1 measurable lesion is confirmed by the lesion assessment at baseline; an evaluable lesion is defined as more than 1.5 cm in greatest dimension and can be followed by imaging.
3. Relapsed or refractory disease after receiving ≥1 prior systemic therapy with antitumor agent(s) and there is no other available treatment which can be considered appropriate for patients. Systemic therapy is defined as frontline chemotherapy or immunotherapy administered systemically.
4. Male or female, age 20 years or older
5. ECOG Performance Status of 0-2
6. Life expectancy of greater than 3 months
7. Meeting the following laboratory criteria for screening:

   1. Absolute Neutrophil Count >1500/µL independent of growth factor support within 7 days of starting the study drug
   2. Platelets >75,000/µL independent of transfusion within 14 days of starting the study drug
   3. Hgb >8 g/dL independent of transfusion within 14 days of starting the study drug
   4. Serum creatinine < 1.5 X ULN
   5. Serum aspartate aminotransferase/glutamyl oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/glutamyl pyruvic transaminase (ALT/SGPT) less than or equal to 3 X ULN
   6. Serum Bilirubin less than or equal to 1.5 X ULN
8. Negative serum pregnancy test for females of childbearing (reproductive) potential. Female patients of child bearing potential must use an effective method of birth control (e.g., hormonal contraceptive, intrauterine device, diaphragm with spermicide or condom with spermicide) during treatment period and 1 month thereafter. Males must use an effective method of birth control (2 barrier methods) during treatment period and 3 months thereafter.

   Note: Female patients will be considered to be women of childbearing potential unless having undergone permanent contraception or postmenopausal. Postmenopausal is defined as at least 12 months without menses with no other medical reasons (e.g., chemical menopause because of treatment with anti-malignant tumor agents)
9. Signed informed consent

Exclusion Criteria:

1. Patients in whom central nervous system lymphoma is recognized during screening (if suspected clinically, imaging study should be performed to confirm)
2. Male patients with QTcF > 450 msec at screening, female patients with QTcF > 470 msec at screening or patients with congenital long QT syndrome, clinically significant arrhythmia, history of congestive heart failure (New York Heart Association Class III or IV) or acute myocardial infarction within 6 months of starting the study drug
3. Patients with known hypersensitivity to benzamide class of compounds or any of the components of HBI-8000 tablets, and patients with prior exposure of HBI-8000
4. Patients with a history of second malignancy other than disease under study. The exceptions are disease that has been treated with curative intent with no evidence of recurrence in past 2 years including:

   1. Basal cell carcinoma of the skin
   2. Squamous cell carcinoma of the skin
   3. Cervical carcinoma in situ
   4. Carcinoma in situ of the breast
   5. An incidental histological finding of prostate carcinoma (TNM stage T1a or T1b)
   6. Early-stage gastric cancer treated with endoscopic mucosal resection or endoscopic submucosal dissection
   7. Thyroid cancer with differentiated histology (e.g. papillary) treated with curative intent
5. Autologous stem cell transplantation within 12 weeks (84 days) of starting the study drug
6. History of allogeneic stem cell transplantation
7. Organ transplantation recipients except autologous hematopoietic stem cell transplantation
8. Uncontrolled inter-current infection
9. Hepatitis B surface antigen-positive, or hepatitis C virus antibody positive. In case hepatitis B core antibody and/or hepatitis B surface antibody is positive even if hepatitis B surface antigen-negative, a hepatitis B virus DNA test (real-time PCR measurement) should be performed and if positive, the patient should be excluded from study
10. Any history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
11. Uncontrolled diabetes mellitus, hypertension, endocrine disorder, bleeding disorder
12. Major surgery or radiation therapy within 28 days of starting the study drug
13. Receiving investigational agents or anti-cancer therapy, within 28 days, nitrosourea or mitomycin C within 42 days of starting the study drug
14. Receiving antibody therapy for PTCL within 12 weeks of starting the study drug
15. Women who are breastfeeding or women who are not willing to stop breastfeeding during study treatment period and for 30 days after the last dose of study drug
16. Potential for non-compliance or at increased risk based on investigator's judgement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-11; Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Lee, MD, Study Chair — HUYABIO International, LLC.
Locations (23):
- Japan (18):
  - Akita
  - Bunkyōku
  - Chūōku
  - Fukuoka
  - Isehara
  - Kagoshima
  - Kobe
  - Kōtoku
  - Kumamoto
  - Kyoto
  - Maebashi
  - Nagoya
  - Okayama
  - Ōmura
  - Sapporo
  - Sayama
  - Suita
  - Yamagata
- South Korea (5):
  - Busan
  - Goyang-si
  - Incheon
  - Seongnam-si
  - Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rai S, Kim WS, Ando K, Choi I, Izutsu K, Tsukamoto N, Yokoyama M, Tsukasaki K, Kuroda J, Ando J, Hidaka M, Koh Y, Shibayama H, Uchida T, Yang DH, Ishitsuka K, Ishizawa K, Kim JS, Lee HG, Minami H, Eom HS, Kurosawa M, Lee JH, Lee JS, Lee WS, Nagai H, Shindo T, Yoon DH, Yoshida S, Gillings M, Onogi H, Tobinai K. Oral HDAC inhibitor tucidinostat in patients with relapsed or refractory peripheral T-cell lymphoma: phase IIb results. Haematologica. 2023 Mar 1;108(3):811-821. doi: 10.3324/haematol.2022.280996. PMID 36200417

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HBI-8000
Started | 55
Completed | 3
Not Completed | 52
Not completed — Adverse Event | 18
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 1
Not completed — Disease Progression | 27

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one dose of HBI-8000.
Arm/Group | HBI-8000
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 55
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 16
  Japan | 39

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Tumor assessment was performed every 8 weeks until disease progression. Objective response rate was defined as the percentage of patients who achieved a complete response (CR) or a partial response (PR) according to International Workshop Response Criteria (IWC) 2014 criteria and assessed by an Independent Overall Efficacy Review Committee (IOERC).
  CR: Target nodes/nodal masses must regress to <1.5 cm in longest transverse diameter of a lesion (LDi), no extralymphatic sites of disease, nonmeasured lesion is absent, disappearance of spleen or liver enlargement, no new lesions, no bone marrow (BM) involvement.
  PR: ≥50% decrease in sum of the product of the perpendicular diameters for multiple lesions (SPD) of up to 6 target measurable nodes and extranodal sites, nonmeasured lesions is absent/normal, regressed, but no increase, spleen must have regressed by >50% in length beyond normal, no new lesions.
Time Frame: Up to approximately 47 months.
Population: The per-protocol analysis set (PPS) included subjects meeting all eligibility criteria who have completed Cycle 1 treatment. For subjects who developed clinical PD and discontinued study treatment during Cycle 1 without significant deviation from protocol, they will be included in the PPS. It should be noted that the PPS includes subjects who discontinued within Cycle 1 due to clinical PD without imaging studies to assess disease status.
Measure: Count of Participants; unit: Participants
Groups:
- HBI-8000: HBI-8000 tablets
Arm/Group | HBI-8000
Number analyzed (Participants) | 46
Participants | 21

2. Secondary Outcome: Objective Response Rate by Disease Subtype
Description: Tumor assessment was performed every 8 weeks until disease progression. Objective response rate was defined as the percentage of patients who achieved a CR or a PR according to IWC 2014 criteria and assessed by an IOERC.
  CR: Target nodes/nodal masses must regress to <1.5 cm in LDi, no extralymphatic sites of disease, nonmeasured lesion is absent, disappearance of spleen or liver enlargement, no new lesions, no BM involvement.
  PR: ≥50% decrease in SPD of up to 6 target measurable nodes and extranodal sites, nonmeasured lesions is absent/normal, regressed, but no increase, spleen must have regressed by >50% in length beyond normal, no new lesions.
  Disease subtype (PTCL-NOS, AITL, ALCL, ALK, EATL) was assessed by Central Pathology Review (CPR).
Time Frame: Up to approximately 47 months.
Population: PPS [Per Protocol Set]
Measure: Count of Participants; unit: Participants
Groups:
- PTCL-NOS: PTCL Not Otherwise Specified
- AITL: Angioimmunoblastic T-cell lymphoma
- ALCL, ALK-: Anaplastic Large-cell Lymphoma, ALK-
- EATL: Enteropathy-associated T-cell lymphoma
Arm/Group | PTCL-NOS | AITL | ALCL, ALK- | EATL
Number analyzed (Participants) | 34 | 8 | 3 | 1
Participants | 12 | 7 | 1 | 1

3. Secondary Outcome: Median Duration of Progression-free Survival (PFS)
Description: PFS was defined as the duration from the date of the first study drug dose to the disease progression or death, whichever occurs first. PD was defined using the IWC 2014 criteria, as any new lesion or an individual node/lesion must be abnormal with: "LDi >1.5 cm" and "increase by 50% from perpendicular diameters nadir" and "an increase in LDi or shortest axis perpendicular to the LDi from nadir, 0.5 cm for lesions <2 cm or 1.0 cm for lesions >2 cm".
Time Frame: Up to approximately 47 months.
Population: PPS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HBI-8000
Number analyzed (Participants) | 46
Months | 5.5 [2.9 to 24.0]

4. Secondary Outcome: Median Duration of Response (DOR)
Description: DOR was defined as the duration of response from first response (CR/PR) to disease progression or death, whichever occurs first. CR or PR according to the IWC 2014 criteria was assessed by an IOERC.
Time Frame: Up to approximately 47 months.
Population: Subjects who achieved PR or CR in the PPS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HBI-8000
Number analyzed (Participants) | 21
Months | 25.7 [5.4 to NA] — Not estimable due to the low number of events

5. Secondary Outcome: Safety Evaluated as Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v.4.0
Description: Safety evaluated as number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
  From date of first study drug to 30±3 days after the last dosing of the study drug or before the initiation of new cancer treatment.
Time Frame: Up to approximately 44 months.
Population: Safety analysis set (SAF) includes all subjects who received at least one dose of HBI 8000.
Measure: Count of Participants; unit: Participants
Arm/Group | HBI-8000
Number analyzed (Participants) | 55
Participants | 51

6. Other Pre Specified Outcome: Median Duration of Overall Survival (OS)
Description: Overall survival is defined as the duration from the first dose of study medication to death from any cause.
Time Frame: Up to approximately 55 months.
Population: PPS - Per Protocol Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HBI-8000
Number analyzed (Participants) | 46
Months | 33.6 [16.5 to NA] — Not estimable due to the low number of events

7. Other Pre Specified Outcome: Pharmacokinetics (Cmax-selected Sites)
Description: Maximum observed plasma concentration (ng/mL), obtained directly from the observed concentration versus time data. Calculated for the C1D1 and C2D1 doses.
Time Frame: 0 (predose) up to 72 hours postdose on C1D1 and 0 (predose) up to 4 hours postdose on C2D1
Population: PK population includes all subjects, at the selected sites in Japan and all sites in South Korea, who have pretreatment baseline and at least 1 blood sample on study providing PK data for HBI-8000.
Measure: Median (Full Range); unit: ng/mL
Groups:
- C1D1: PK Sampling on C1D1
- C2D1: PK Sampling on C2D1
Arm/Group | C1D1 | C2D1
Number analyzed (Participants) | 26 | 8
ng/mL | 220 [71.9 to 650] | 254 [118 to 483]

8. Other Pre Specified Outcome: Pharmacokinetics AUC (0-INF)
Description: Area under the plasma concentration time curve from zero (predose) extrapolated to infinity (ng*h/mL) (Day 1 only), calculated by linear up/log down trapezoidal summation and extrapolated to infinity by addition of the last quantifiable concentration (Clast) divided by the apparent terminal rate constant (λz): AUC(0-last) + Clast/λz. Calculated for the C1D1 dose only.
Time Frame: 0 (predose) up to 72 hours postdose on C1D1
Population: as for outcome 7
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | C1D1
Number analyzed (Participants) | 26
ng*h/mL | 5330 [2230 to 9110]

9. Other Pre Specified Outcome: Pharmacokinetics AUC (0-tau)
Description: Area under the plasma concentration time curve over the dosing interval tau (ng*h/mL), calculated by linear up/log down trapezoidal summation. Calculated for the C1D1 dose only. Actual elapsed sampling time at tau and the corresponding plasma concentration was used in the calculation of this parameter. If concentrations fall to BLQ before or at tau, AUCall (area under the plasma concentration time curve from zero [predose] to the time of the last observation within the dosing interval, calculated by linear up/log down trapezoidal summation) was used as the estimate of this parameter.
Time Frame: 0 (predose) up to 72 hours postdose on C1D1
Population: as for outcome 7
Measure: Median (Full Range); unit: ng*h/mL
Groups:
- C1D1: PK Sampling C1D1
Arm/Group | C1D1
Number analyzed (Participants) | 26
ng*h/mL | 4740 [2130 to 8630]

10. Other Pre Specified Outcome: t 1/2
Description: Apparent terminal half-life (h), calculated as (ln 2)/λz. Calculated for the C1D1 dose only.
Time Frame: 0 (predose) up to 72 hours postdose on C1D1
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | C1D1
Number analyzed (Participants) | 26
hour | 17.7 [14.3 to 25.5]

ADVERSE EVENTS:
Time Frame: From date of the first study drug to 30 ± 3 days after the last dosing of the study drug or before the initiation of new cancer treatment, an average of around 7 months.
Description: Other (Not Including Serious) Adverse Events: Adverse events include Serious Adverse Events.
Arm/Group | HBI-8000
All-Cause Mortality (participants affected / at risk) | 1/55
Serious Adverse Events (participants affected / at risk) | 15/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBI-8000 (N=55)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBI-8000 (N=55)
Anaemia (Blood and lymphatic system disorders) | 19 (19)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (16)
Neutropenia (Blood and lymphatic system disorders) | 11 (11)
Leukopenia (Blood and lymphatic system disorders) | 6 (6)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Palpitations (Cardiac disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 19 (19)
Nausea (Gastrointestinal disorders) | 12 (12)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Toothache (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Pyrexia (General disorders) | 13 (13)
Malaise (General disorders) | 9 (9)
Fatigue (General disorders) | 6 (6)
Oedema peripheral (General disorders) | 5 (5)
Nasopharyngitis (Infections and infestations) | 5 (5)
Pharyngitis (Infections and infestations) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Bronchitis (Infections and infestations) | 3 (3)
Platelet count decreased (Investigations) | 31 (31)
Neutrophil count decreased (Investigations) | 21 (21)
White blood cell count decreased (Investigations) | 19 (19)
Lymphocyte count decreased (Investigations) | 12 (12)
Blood alkaline phosphatase increased (Investigations) | 8 (8)
Gamma-glutamyltransferase increased (Investigations) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 7 (7)
Weight decreased (Investigations) | 7 (7)
Alanine aminotransferase increased (Investigations) | 6 (6)
Electrocardiogram QT prolonged (Investigations) | 5 (5)
C-reactive protein increased (Investigations) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 14 (14)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 7 (7)
Insomnia (Psychiatric disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (5)
Purpura (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HUYABIO International, LLC has agreements with PIs and the agreements restricts the right of the PI to discuss or publish trial results after the trial is completed.

The content of disclosure restriction stated in the agreement is "PI shall obtain sponsor's prior written consent before disclosing the information obtained from this clinical trial to a professional society or other external party."

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT02953652/Prot_SAP_000.pdf